CLINICAL TRIAL: NCT07118007
Title: Assessment of the Benefits of Adapted Physical Activity in Pediatric Hemodialysis Patients-DIALAPA Study
Brief Title: Assessment of the Benefits of Adapted Physical Activity in Pediatric Hemodialysis Patients
Acronym: DIALAPA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL25_0588
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Hemodialysis
Keywords: Hemodialysis; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient requiring hemodialysis for end-stage renal disease (Other): Patient requiring hemodialysis for end-stage renal disease aged 5 to 20 years
  Interventions: Other: adapted physical activity

INTERVENTIONS:
Other: adapted physical activity — adapted physical activity for 30 to 45 minutes twice per week

SUMMARY:
Children, adolescents, and young adults undergoing pediatric hemodialysis often experience functional limitations in daily life. Their level of physical activity is generally lower than that of healthy peers of the same age, due to the lack of sports programs adapted both to their medical conditions and to the constraints of dialysis (notably, having to remain in bed for several hours, several times a week). These limitations affect not only their cardiovascular function but also their quality of life.

Through the implementation of an Adapted Physical Activity (APA) program for dialysis patients, we aim to assess the potential benefits of this approach on muscle strength, functional abilities, cardiovascular health, and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring hemodialysis sessions for end-stage renal disease
* Patient aged between 5 and 20 years
* Patient followed in the pediatric nephrology department at hospital Lyon (HFME : Hôpital Femme Mère Enfant)
* Adult patient or parents/legal guardians informed about the study and having provided written consent for participation
* Patient covered by a social security

Exclusion Criteria:

Medical or surgical contraindications to adapted physical activity.

* Persons deprived of liberty by judicial or administrative decision.
* Persons undergoing psychiatric care.
* Persons admitted to a healthcare or social facility for reasons other than research participation.
* Adults under legal protection measures (curators)
* Persons not affiliated with a social security scheme or beneficiaries of a similar system
* Pregnant women.

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
mass-to-muscle mass ratio between M0 and M6 | Between baseline (M0) and month 6 (M6)
  Change in the mass-to-muscle mass ratio between M0 and M6, measured at the end of the hemodialysis session using bioelectrical impedance analysis.

IPD SHARING:
Plan to Share IPD: No